CLINICAL TRIAL: NCT06153615
Title: Sleeping With Open Eyes: Local Sleep in Idiopathic Hypersomnia
Brief Title: Local Sleep in Idiopathic Hypersomnia
Acronym: SL-HIP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: APHP230749
Record Dates: First submitted 2023-09-29; First posted 2023-12-01 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Idiopathic Hypersomnia
Keywords: Idiopathic Hypersomnia; Narcolepsia type 1
MeSH Terms: conditions — Idiopathic Hypersomnia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Idiopathic Hypersomnia (Experimental)
  Interventions: Other: EEG (64 electrodes); Other: Cognitive task (SART); Other: Pupillometry and eye tracking; Other: Thoracoabdominal belts
- Narcolepsy type 1 (Active Comparator)
  Interventions: Other: EEG (64 electrodes); Other: Cognitive task (SART); Other: Pupillometry and eye tracking; Other: Thoracoabdominal belts
- Healthy subject (Active Comparator)
  Interventions: Other: EEG (64 electrodes); Other: Cognitive task (SART); Other: Pupillometry and eye tracking; Other: Thoracoabdominal belts

INTERVENTIONS:
Other: EEG (64 electrodes) — EEG recording while awake, at rest then during an attentional cognitive test
Other: Cognitive task (SART) — Sustained attention go-no-go task (press a button each time a number is presented on a screen (1/second) except when the 3 appears) Assessment of mental status approximately every 45 seconds (task focus, mind wandering, mental blank, and sleepiness status)
Other: Pupillometry and eye tracking — Study of pupil size and gaze path during the cognitive test (correlated with alertness)
Other: Thoracoabdominal belts — Abdominal and thoracic belts (used in all nocturnal polysomnographic recordings) for respiratory movement studies (correlated with sleepiness)

SUMMARY:
Idiopathic hypersomnia (IH) is a rare and poorly studied disease characterized by excessive daytime sleepiness different from that of narcolepsy (sleep drunkness non-recuperative naps and nocturnal blackout). Local sleep is a recent concept, proposing a local regulation of the sleep-wake state, characterized by slow waves (SW) restricted to certain regions of a globally awake brain. The investigators are going to investigate whether local sleep could explain the sleepiness of these patients better than the global occurrence of sleep which are not very frequent during daytime tests in IH.

The investigators propose to look for local sleep through the detection of local slow waves in the EEG of resting wakefulness and during an attentional task in people with IH compared to people with NT1 (sleepy, but with a different type of sleepiness from IH, more abrupt and including REM sleep) and non sleepy people.

DETAILED DESCRIPTION:
Local sleep is a recent concept, suggesting a local regulation of the sleep-wake state, characterized for example in wakefulness by slow waves restricted to certain regions of a globally awake brain, correlating with modifications of mental experience and behavior. Although the phenomenon of local sleep has been demonstrated following acute sleep deprivation, its importance in explaining attentional fluctuations during a normal day is only beginning to be investigated. Moreover, inter-individual variations remain unexplored. The investigators propose to study in EEG (64 electrodes) the occurrence of local sleep in different states of sleepiness, in particular in idiopathic hypersomnia (IH) in comparison to that of narcolepsy type 1 (NT1) and to non-drowsy individuals, both in the resting state and during a sustained attention test (SART). This study will provide a better understanding of intra- (over the course of a day) and inter-individual fluctuations in the local sleep phenomenon potentially involved in this disease and its impact on cognition.

Anticipated number of participants:

60 including:

* 20 people with idiopathic hypersomnia
* 20 people with type 1 narcolepsy
* 20 people with no previous history

Practical procedure:

Single visit: presence from 9:30 am to 3:30 pm

* General questionnaire on sleep habits and symptoms.
* Equipment: EEG 32 electrodes, EOG, ECG, eye tracker and thoracoabdominal belts.
* Morning and afternoon recording: 10 minutes in resting state, 60 minutes of digital SART (go-no-go test in front of a screen, with intermittent evaluation of mental state), then 10 minutes of rest.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria :

* Healthy subjects and people with IH and NT1:

  ->18 years old, of both sexes, without legal protection.
  * Affiliated to the French social security system
  * Signature of free and informed consent
  * Fluency in spoken and written French
* Specific to people with IH:

  -Diagnosis of IH according to the ICSD-3, already made in the sleep pathology department of the Pitié after a specialized medical interview and a standardized 48h assessment (Night 1+TILE+Night 2+two naps): Sleep time > 660 min or TILE latency <8 min, <2 SOREMPs.
* Specific to people with NT1:

  * Diagnosis of narcolepsy type 1 according to the ICSD-3, already made in the sleep pathology department of the Pitié after a specialized medical interview and a standardized 48h workup (Night 1+TILE+Night 2+two naps) and sometimes a lumbar puncture: hypocretin <110 pmol/L in CSF or cataplexy and TILE latency <8 min, >1 SOREMP.

Exclusion Criteria:

* Shift or night work
* Sleep debt on the day of the recording (questioning and sleep diary one week before the recording)
* Other sleep pathology causing daytime sleepiness (sleep apnea, insomnia, parasomnia for example)
* Cerebral neurological pathology
* Depressive episode
* Any psychotropic treatment modifying the EEG structure
* Failure to wean from arousing treatment on the day of the test.
* Inability to travel by transport or to be transported by a relative on the day of the recording.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-12 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
local sleep topography | At enrollment visit
  Density and topography of local sleep through the detection of local slow waves (SW) during resting wakefulness and during a daytime attentional test in IH, narcolepsy and healthy subjects

SECONDARY OUTCOMES:
Daytime dynamics of local sleep | At enrollment visit
  Density and topography of local sleep through the detection of local slow waves at two times of the day.
behavioral implications of local sleep | At enrollment visit
  Correlation of slow wave characteristics to mental experience and performance (reaction time, omission, impulsivity) during the sustained attention task.
correlation between local sleep and behavioral marker of alertness | At enrollment visit
  Correlation of pupillometric and eye tracking measurements, respiratory and heart rate parameters (assessments correlated to the state of alertness) to the different measured parameters

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle Arnulf, MD, PhD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pitié Salpêtrière, Paris, France

IPD SHARING:
Plan to Share IPD: No
The data will be confidential until their publication in a peer reviewed journal. Sharing will be feasible after, in case of reasonable request to the PI.